CLINICAL TRIAL: NCT02888964
Title: A Study to Assess Efficacy and Safety of Pioglitazone as Add-On Therapy to Imatinib Mesylate in CP-CML Patients in Major Molecular Response
Brief Title: Pioglityazone and Imatinib for CML Patients
Acronym: ACTIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Philippe ROUSSELOT, Study Coordinator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/37_ACTIM
Record Dates: First submitted 2016-08-19; First posted 2016-09-05 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACTOS treatment (Experimental): Imatinib mesylate at the same daily dose and pioglitazone as add-on therapy at 30 mg/d during 2 months and then 45 mg/d in the absence of serious adverse events
  Interventions: Drug: Add-on therapy

INTERVENTIONS:
Drug: Add-on therapy — Pioglitazone therapy

SUMMARY:
This project is a Phase II clinical trial that aims at evaluating efficacy and tolerance of the combination of pioglitazone (Actos®) and imatinib mesylate (STI571, CGP57148, Gleevec®) in patients with Chronic Myelogenous Leukemia (CML) in stable major molecular response (i.e. a BCRABL/ABL ratio assessed by RTQ-PCR equal to or lower than 0.1% according to the European Leukemia Net recommendations) after at least 2 years of therapy with imatinib.

Imatinib mesylate (Gleevec®) is the gold standard for the treatment of CML in chronic phase (O Brian et al. 2003, Druker et al. 2006). Despite a high efficacy of the drug, CML is not eradicated by imatinib alone in almost any of the patients.

Treatment discontinuation in patients treated by imatinib and in complete molecular remission for more than 2 years yield molecular relapses within 6 months in half of the patients,indicating the persistence of CML progenitor cells. STAT5 expression is required for CML stem cell engraftment and expansion in mouse models. STAT5 is the target of the dysregulated activity of BCR-ABL in CML.

Recently, Stephane Prost et al. demonstrated that PPAR-γ is a negative regulator of STAT5A and STAT5B gene expression. Data obtained suggest that PPAR-γ agonists may have potential therapeutic value in reversing myeloproliferative disorders. On the basis of our preclinical studies, we went ahead and administered pioglitazone to one patient who suffered from both diabetes type II and CML with residual disease after continuous treatment with Gleevec. The amount of BCR-ABL transcript detected by QPCR decreased dramatically during the first 3 months of combined (Gleevec + ACTOS) therapy to become undetectable thereafter until 9 months post-treatment, the latest time point assessed. This striking anecdotal result now forms the rationale for filing this formal Phase II clinical trial application.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18y or more
2. Signed informed consent
3. Patient with Philadelphia chromosome positive chronic phase CML and M BCR-ABL transcript positivity
4. Treatment with imatinib for more than 2 years
5. No dose modification of imatinib within the last 3 months
6. Complete cytogenetic response on the last cytogenetic analysis within the last 12 months
7. Major molecular remission without complete molecular remission
8. ECOG grade 0 to 2
9. SGOT et SGPT ≤ 2.5 N
10. Bilirubin in serum ≤ 1.5 N
11. Women of childbearing potential (WOCBP) must be using an adequate method of contraception

Exclusion Criteria:

1. Participation in another clinical trial with any investigative drug within 30 days prior to study enrollment
2. Prior history of hematopoietic stem cell transplantation (autologous or allogenic)
3. Patient requiring anti-diabetic medication
4. Cardiovascular disease:

   * Stage I to IV congestive heart failure (CHF) as determined by the New York Heart Association (NYHA) classification system for heart failure
   * Myocardial infarction within the previous 6 months
   * Symptomatic cardiac arrhythmia requiring treatment
5. Grade III or IV fluid retention
6. Known osteoporosis with therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The rate of patients achieving a complete molecular response (Sensitivity 10-5 or Bcr Abl/Abl ratio < 0.001 %) 24 weeks after the initiation of pioglitazone, confirmed on by a second determination 2 months later. | 26 weeks

SECONDARY OUTCOMES:
Adverse events | 5 years
Duration of the complete molecular response | 5 years
The rate of patients achieving a complete molecular response (Sensitivity 10-5 or Bcr-Abl/Abl ratio < 0.001 %) | 14 months
Survival | 5 years
Progression free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rousselot Philippe, MD, Principal Investigator — CH Versailles
Locations (9):
- France (9):
  - CHR Annecy, Annecy
  - Institut Bergonié, Bordeaux
  - CH Versailles, Le Chesnay
  - CHU Lille, Lille
  - IPC, Marseille
  - CHU archet 1, Nice
  - St Louis, Paris
  - CHU Poitiers, Poitiers
  - CHU Purpan, Toulouse